CLINICAL TRIAL: NCT03500874
Title: Adjuvant Systemic Chemotherapy With or Without Hepatic Arterial Infusion Using Floxuridine in Patients Following Colorectal Cancer Liver Metastases Resection
Brief Title: Adjuvant Systemic Chemotherapy With or Without HAI-FUDR in Patients With Resected CRLM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely due to FUDR production halt in China
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAI-CRCLM-ADJUVANT
Record Dates: First submitted 2018-04-08; First posted 2018-04-18 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Liver Metastases; HAI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Floxuridine; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAI group (Experimental): Patients will receive systemic chemotherapy on days 1 and 15 using either of the following regimens: mFOLFOX6 (Oxaliplatin 85 mg/m2; Leucovorin 200mg/m2; followed by an infusion of 5-fluorouracil 2.4 g/m2 administered over 46 hours) or mFOLFIRI (Irinotecan 180mg/m2; Leucovorin 200mg/m2; followed by an infusion of 5-fluorouracil 2.4 g/m2 administered over 46 hours) For HAI, FUDR was administered as a continuous infusion of 0.12 mg/kg/day over 14 days via the HAI pump, along with dexamethasone 20 mg, and normal saline was used to fill up the 300ml pump reservoir.
  Interventions: Drug: FUDR; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5FU; Drug: Irinotecan
- Non-HAI group (Active Comparator): Patients will receive systemic chemotherapy on days 1 and 15 using either of the following regimens: mFOLFOX6 (oxalipatin 85 mg/m2 infusion for 3 h, Leucovorin 200 mg/m2 for 3 h and 5-FU 2,400 mg/m2 continuous infusion for 46 h) or mFOLFIRI (Irinotecan 180mg/m2; Leucovorin 200mg/m2; 5-FU 2,400 mg/m2 continuous infusion for 46 h).
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5FU; Drug: Irinotecan

INTERVENTIONS:
Drug: FUDR — Floxuridine(FUDR) 0.12 mg/kg/day，on Day 1-14 through the HAI pump.
  Other Names: Floxuridine
  Arms: HAI group
Drug: Oxaliplatin — Oxaliplatin 180 mg/m2 IV over 90 minutes on Day 1, 15.
  Other Names: Xaliplatin
Drug: Leucovorin — Leucovorin 200mg/m2 ivd over 2 hours on Day 1
  Other Names: Folinic Acid
Drug: 5FU — 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1.
  Other Names: 5-Fluorouracil
Drug: Irinotecan — Irinotecan 180mg/m2
  Other Names: CPT-11

SUMMARY:
HARVEST is an investigator-initiated prospective randomized controlled study comparing adjuvant intravenous systemic chemotherapy with or without HAI- floxuridine (FUDR) in CRC patients post-liver metastasectomy.

DETAILED DESCRIPTION:
Numerous retrospective studies have indicated a positive synergistic effect of combining adjuvant oxaliplatin/irinotecan-based doublet systemic chemotherapy and hepatic arterial infusion (HAI) for colorectal cancer (CRC) patients following colorectal cancer liver metastases (CRLM) resection. However, this strategy has not been evaluated prospectively to date. HARVEST is an investigator-initiated prospective randomized controlled study comparing adjuvant intravenous systemic chemotherapy with or without HAI- floxuridine (FUDR) in CRC patients post-liver metastasectomy.

ELIGIBILITY:
Inclusion Criteria:

1. The primary lesion has undergone or is capable of radical resection, and liver metastases can undergo R0/R1 resection (including intraoperative interventional ablation therapy), and postoperative achievement of no evidence of disease (NED).
2. Histologically confirmed colorectal adenocarcinoma
3. Radiologically or pathologically confirmed diagnosis of colorectal liver metastasis
4. No previous surgery, interventional ablation, hepatic arterial infusion (HAI), radiotherapy, or transarterial chemoembolization (TACE) for liver metastases.
5. CT, MRI, or PET/CT (if necessary) confirmed no extrahepatic metastasis.
6. Normal hematologic function (platelets > 90×10^9/L; white blood cells > 3×10^9/L; neutrophils > 1.5×10^9/L).
7. No ascites, normal coagulation function, albumin ≥ 35g/L.
8. Liver function graded as Child-Pugh class A.
9. Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), transaminases ≤ 5 times ULN, alkaline phosphatase ≤ 2.5 ULN.
10. Serum creatinine below the upper limit of normal (ULN), or calculated creatinine clearance > 50ml/min (using Cockcroft-Gault formula).
11. ECOG performance status of 0-2
12. Life expectancy ≥ 3 months
13. Patients have provided a signed Informed Consent Form
14. Willing and able to undergo follow-up until death or the end of the study or study termination.

Exclusion Criteria:

1. Have had any extrahepatic metastasis after being diagnosed with colorectal cancer.
2. Previous surgery, interventional ablation, hepatic arterial infusion (HAI), radiotherapy, or transarterial chemoembolization (TACE) for liver metastases.
3. Liver metastases intended for interventional ablation treatment only.
4. Presence of hepatic artery vascular variation identified by CTA examination, making HAI implantation unsuitable.
5. Severe arterial embolism or ascites.
6. Bleeding tendency or coagulation disorders.
7. Hypertensive crisis or hypertensive encephalopathy.
8. Severe uncontrollable systemic complications such as infection or diabetes.
9. Clinically significant cardiovascular diseases such as cerebrovascular accidents (in the last 6 months before enrollment), myocardial infarction (in the last 6 months before enrollment), uncontrolled hypertension despite appropriate drug treatment, unstable angina, congestive heart failure (NYHA 2-4), and arrhythmias requiring medication.
10. History of or physical examination indicating central nervous system diseases (such as primary brain tumors, uncontrollable epilepsy, any brain metastasis, or history of stroke).
11. Had any other malignant tumors in the past 5 years (excluding basal cell carcinoma and/or cervical carcinoma in situ after radical surgery).
12. Received any investigational drug treatment in the last 28 days before the study.
13. Any residual toxicity from previous chemotherapy (excluding alopecia), such as peripheral neuropathy ≥ NCI CTC v3.0 grade 2, makes the use of a treatment regimen containing oxaliplatin not considered.
14. Allergic to any drugs in the study.
15. Pregnant or lactating women who are not using or refuse to use effective non-hormonal contraception (intrauterine device, barrier contraception combined with spermicidal gel, or sterilization) in women of childbearing age (last menstrual period < 2 years ago) or fertile men who cannot or do not wish to comply with the study protocol.
16. Presence of any other diseases, functional impairment due to metastatic lesions, or suspicious findings in the physical examination suggesting contraindications to the use of the investigational drug or placing the patient at a high risk of treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
3 Year Relapse Free Survival Rate | up to 36 months
  Calculated from the time of liver metastasectomy to the time of recurrence or death, whichever came first or censored at the date of the last follow-up for recurrence-free patients that were still alive

SECONDARY OUTCOMES:
Overall Survival | up to 5 years
  From date of randomization until the date of death from any cause, assessed up to 5 years
Treatment-related adverse events | Up to 36 months
  Number of patients with adverse events and severity measured according to the NCI CTC 3.0 criteria
Liver-specific RFS | Up to 36 months
  Measure of the time period during which a patient remains free from the recurrence of liver-related events

OTHER OUTCOMES:
Serum ctDNA methylation levels | Up to 5 years
  The methylation status of blood ctDNA at a specific time point (e.g., postoperatively) was considered positive if either of the two markers (SEPT9 and NPY) yielded results above zero. Conversely, it was deemed negative if both markers showed an absence of methylation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol

REFERENCES:
- [Derived] Wang DS, Pat Fong W, Wen L, Cai YY, Ren C, Wu XJ, Zhang TQ, Cao F, Zuo MX, Li BK, Zheng Y, Li LR, Chen G, Ding PR, Lu ZH, Zhang RX, Yuan YF, Pan ZZ, Li YH. Safety and efficacy of adjuvant FOLFOX/FOLFIRI with versus without hepatic arterial infusion of floxuridine in patients following colorectal cancer liver metastasectomy (HARVEST trial): A randomized controlled trial. Eur J Cancer. 2025 Jan;214:115154. doi: 10.1016/j.ejca.2024.115154. Epub 2024 Nov 30. PMID 39644535